CLINICAL TRIAL: NCT01590108
Title: The Apelin-APJ System in Idiopathic Pulmonary Arterial Hypertension and Healthy Volunteers; Tissue Location and Cardiopulmonary Response.
Brief Title: The Study of Apelin-APJ System on Pulmonary Hypertension Patients and Healthy Subjects
Acronym: EXAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11/LO/2063
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
Keywords: Idiopathic Pulmonary Arterial Hypertension; IPAH; Apelin; APJ receptor
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — apelin 13, Pyr(1)-; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apelin (Experimental): Subject will perform cardiopulmonary exercise testing and receive (Pyr1)apelin-13 intravenously.
  Interventions: Drug: (Pyr1)apelin-13
- Control (Placebo Comparator): Subject will take cardiopulmonary exercise testing with receive placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: (Pyr1)apelin-13 — (Pyr1)apelin-13 will be infused at 30 nanomol/min intravenously. This dose has been used in healthy volunteer and patients groups
  Arms: Apelin
Drug: Saline — Saline
  Arms: Control

SUMMARY:
The purpose of this study is to

* Determine blood peptide levels and investigate any tissue gradients of apelin in patients with idiopathic pulmonary arterial hypertension and healthy volunteers.
* Evaluate the effect of exogenous apelin infusion on exercise performance in healthy volunteers and patients with idiopathic pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Idiopathic pulmonary arterial hypertension remains an enigma for physician in both diagnosis and treatment. Existing biomarkers, tissue characteristics and definite treatment are restricted. There are many evidences suggested that Apelin-APJ system associated with Idiopathic Pulmonary Arterial Hypertension (IPAH). A comprehensive characterise circulating peptide levels and investigate any tissue gradients of apelin in patients with idiopathic pulmonary arterial hypertension and healthy volunteers might provide important information about pathophysiologic process and diagnostic marker. In addition, first time human study to assessment the effect of exogenous apelin infusion on exercise performance in healthy volunteers and patients with idiopathic pulmonary arterial hypertension is essential to confirm whether the relevance between animal models and clinical subjects.

ELIGIBILITY:
Inclusion Criteria for Control group:

* Structurally normal heart by 2D Echocardiography
* Pulmonary artery pressure < 25mmHg
* Tricuspid velocity < 2.5ms-1

Inclusion Criteria for Treatment group:

* Clinical diagnosis of Pulmonary arterial hypertension that is idiopathic, associated with anorexigens associated with connective tissue disease or familial
* Able to give informed consent
* Mean pulmonary artery pressure > 25mmHg, pulmonary capillary wedge pressure < 15mmHg, with normal or reduced cardiac output.

Exclusion Criteria for ALL group:

* Bleeding diathesis (PT > 14 sec to aPTT > 40 sec)
* Pregnancy, or women of child bearing potential not on adequate contraception
* Renal or hepatic failure
* Severe valvular heart disease
* Left ventricular dysfunction (LVEF < 40)
* Chronic lung disease
* Malignant arrhythmias
* Chronic thromboembolic disease

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Effect of Apelin infusion on cardiopulmonary performance in healthy volunteers and patient with idiopathic pulmonary hypertension | 6 months
  Characterise circulating peptide levels and investigate any tissue gradients of apelin in patients with idiopathic pulmonary arterial hypertension and healthy volunteers.
  Assess the effect of exogenous apelin infusion on exercise performance in healthy volunteers and patients with idiopathic pulmonary arterial hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Sebastian Howard, DPhil, Principal Investigator — Imperial College NHS Trust; Gareth D Barnes, MBChB, Study Director — Imperial College NHS trust
Locations (2):
- United Kingdom (2):
  - Hammersmith Hospital, Imperial College London, London
  - Imperial College Healthcare NHS Trust, London